CLINICAL TRIAL: NCT00114764
Title: A Multicentre, Double-Blind, Randomised Phase 2 Trial Comparing Pegfilgrastim With Filgrastim as an Adjunct to Chemotherapy for Acute Myeloid Leukaemia (AML)
Brief Title: Trial Comparing Pegfilgrastim With Filgrastim as an Adjunct to Chemotherapy for Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20020163
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Myeloid Leukemia
Keywords: Acute myeloid leukaemia; Pegfilgrastim; Neulasta®; Neutropenia; Induction chemotherapy; Consolidation
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute; Neutropenia | interventions — Filgrastim; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- pegfilgrastim (Experimental): Pegfilgrastim given once after induction chemotherapy
  Interventions: Drug: pegfilgrastim
- filgrastim (Active Comparator): Filgrastim given daily after induction chemotherapy
  Interventions: Drug: filgrastim

INTERVENTIONS:
Drug: filgrastim — Filgrastim given daily after induction chemotherapy
  Arms: filgrastim
Drug: pegfilgrastim — Pegfilgrastim given once after induction chemotherapy
  Arms: pegfilgrastim

SUMMARY:
The purpose of this study is to determine if a single dose of pegfilgrastim is able to reduce the time of severe neutropenia in patients receiving induction and consolidation myelosuppressive chemotherapy for de novo acute myeloid leukemia similar to filgrastim.

ELIGIBILITY:
Inclusion

* Histologically confirmed de novo AML as evidenced by absence of an antecedent hematologic disease of > 1 months duration, prior chemotherapy, prior radiation therapy or myelodysplastic cytogenetics (as per exclusion criteria)
* Life expectancy, with treatment, > 3 months
* Age > 18 years
* ECOG performance status 0, 1 or 2
* Adequate organ function to receive protocol specified chemotherapy

Exclusion

* Subjects in blast transformation of chronic myeloid leukaemia (CML)
* Patients with secondary AML (Received previous chemotherapy or radiotherapy)
* Previous treatment for AML
* Patients with AML FAB type M3 (Acute Promyelocytic Leukemia, APL) or M7
* High risk (Unfavourable) cytogenetics [(-5/del(5q), -7/del(7q), t(8;21) with del (9q) or complex karyotype, inv(3q), abn 11q23, 20q, 21q, del(9q), t(6;9), t(9;22), abn 17p, complex karyotypes(>3 abnormalities)]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-03; Primary Completion 2004-04 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Time to recover from severe neutropenia (ANC less that 0.5 X 10^9/L in chemotherapy Induction 1. | Induction cycle 1

SECONDARY OUTCOMES:
Duration of severe neutropenia during induction chemotherapy | Induction cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Sierra J, Szer J, Kassis J, Herrmann R, Lazzarino M, Thomas X, Noga SJ, Baker N, Dansey R, Bosi A. A single dose of pegfilgrastim compared with daily filgrastim for supporting neutrophil recovery in patients treated for low-to-intermediate risk acute myeloid leukemia: results from a randomized, double-blind, phase 2 trial. BMC Cancer. 2008 Jul 10;8:195. doi: 10.1186/1471-2407-8-195. PMID 18616811
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com